CLINICAL TRIAL: NCT03595423
Title: Retrospective Multicentric Study Spanish SPALVALVE: Follow-up to 15 Years of Patients Between 50-65 Years Undergoing Isolated Aortic Valve Replacement. Biological or Mechanical Prostheses
Brief Title: SPAnish Aortic VALVE Multicentric Study
Acronym: SPAVALVE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud (Other)
Responsible Party: Sponsor
Other Study IDs: SPAVALVE
Record Dates: First submitted 2018-07-11; First posted 2018-07-23 (Actual); Last update posted 2018-07-23 (Actual); Status verified 2018-07

CONDITIONS: Survival, Prosthesis; Prosthesis Durability; Valve Heart Disease
Keywords: long-term survival; bioprosthesis
MeSH Terms: conditions — Prosthesis Failure; Heart Valve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bioprosthesis: All patients operated on of isolated AVR with a bioprosthesis implantation between 2000-2015 and age 50-65 years both inclusive.
  Interventions: Procedure: Surgical AVR with bioprosthetic or mechanical prosthesis
- Mechanical prosthesis: All patients operated on of isolated AVR with a Mechanical prosthesis implantation between 2000-2015 and age 50-65 years both inclusive.
  Interventions: Procedure: Surgical AVR with bioprosthetic or mechanical prosthesis

INTERVENTIONS:
Procedure: Surgical AVR with bioprosthetic or mechanical prosthesis — Surgical AVR with bioprosthetic or mechanical prosthesis

SUMMARY:
Currently there is an increase in the use of bioprosthesis worldwide (> 70% according to national data of the Spanish Society of Thoracic and Cardiovascular Surgery). There is conflicting evidence regarding the long-term survival of patients aged 50-65 years with mechanical (M) or biological (B) aortic prostheses. General consensus of greater complications associated with the use of long-life anticoagulation in M and of reoperation in B.

Similar survival with lower MACCE complications in bioprosthesis could reconsider their choice in patients aged 50-65 years, specially in the current TAVI era. The investigators are going to perform a multicentric retrospective observational study (Registry) about 15 year-outcomes Following Bioprosthetic vs Mechanical Isolated Aortic Valve Replacement for Aortic Stenosis in Patients Aged 50 to 65 Years in 30 Cardiovascular Surgery Centers in Spain

DETAILED DESCRIPTION:
Objectives The main objective is to analyze long-term survival (15 years) and major cardiovascular complications (MACE, (early 30-day death, stroke, any prosthesis reoperation, and major bleeding), in patients aged 50-65 years who underwent isolated aortic valve replacement (AVR) due to severe aortic stenosis . Secondary objectives were to analyze the evolution of transprosthetic gradients by echocardiography,, and degree of significant structural degeneration in bioprostheses.

Material and Method: A retrospective analytical study of patients aged 50-65 years who underwent AVR surgery for stenosis between 2000-2015 in 30 centers with a Cardiovascular Surgery Dept. in SPAIN as an inclusion criterion. As exclusion criteria, autonomic change of residence, need for concomitant surgery, previous cardiac interventions and infective endocarditis.

Survival analysis and clinical data records will be performed through the Public Health Care computed medical records , and direct telephone contact with family and / or relatives, in case of doubts. A crude analysis of the data and a posterior analysis by propensity score matching with SPSS or R software will be carried out using a 1: 1 or 2:1 "nearest neighbour" matching protocol based on the Number of total bioprosthesis. A total sample of more than 5000 cases is expected, of which about 1000 would be bioprostheses that would serve as a basis for the pairing. According to previous data(ANDALVALVE STUDY), to find a 4.8% difference in the primary endpoint, two groups of 1025 patients are required for a p = 0.05 and 80% for a bilateral contrast of two independent proportions. Subanalysis will be performed by subgroups of age (50-55 vs. 55-65 years) and another according to the mark of the 2 prostheses of each type most implanted. All statistical analyzes will be two-tailed with an alpha error of 0.05 to consider statistically significant data, and will be reviewed by IBIMA or Private biostatistics. Competing risks analysis will be performed to calculate the cumulative incidence of stroke, reoperation and major bleeding for each prosthesis type.

Conclusions: A positive result (similar survival in group B, with lower complications) could change the current indications of AVR in our environment, allowing the age of indication for bioprostheses in European guidelines to be reduced below 60 years

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 50-65 years who underwent isolated aortic valve replacement (AVR) for severe aortic stenosis from years 2000-2015 both inclusive

Exclusion Criteria:

* Not reported Residency change (unreachable)
* Need of concomitant surgery
* Reoperations
* Infective endocarditis

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 50-65 years who underwent isolated aortic valve replacement (AVR) for severe aortic stenosis from years 2000-2015 both inclusive, with bioprosthesis or mechanical prosthesis implantation
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2018-07-10 (Actual); Primary Completion 2019-03-31 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants alive | From date of surgery until the date of death from any cause, assessed up to 18 years
  Survival since surgery
Late postoperative combined endpoint of 4 Major Adverse Cardiovascular Events (MACE) complications | From date of surgery until the date of first documented MACE (see description) or date of death from any cause, whichever came first, assessed up to 18 years
  Early 30-day Mortality, major bleeding, stroke and need of any prosthesis reoperation

SECONDARY OUTCOMES:
Cumulative incidence of stroke at 15 years between groups | From date of surgery until the date of first documented stroke or date of death from any cause, whichever came first, assessed up to 18 years
  stroke cumulative incidence over time (competing risk analysis)
Cumulative incidence of prosthesis reoperation at 15 years between groups | From date of surgery until the date of first documented reoperation or date of death from any cause, whichever came first, assessed up to 18 years
  reoperation cumulative incidence over time (competing risk analysis)
Cumulative incidence of major bleeding at 15 years between groups | From date of surgery until the date of first documented major bleeding or date of death from any cause, whichever came first, assessed up to 18 years
  major bleeding cumulative incidence over time (competing risk analysis)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Virgen de La Victoria, Málaga, Spain